CLINICAL TRIAL: NCT02913872
Title: Childhood Asthma Management in Primary Care: Implementation Of Exhaled Nitric Oxide and Spirometry Testing
Acronym: CHAMPIONS
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: Aerocrine AB (Industry)
Responsible Party: Sponsor
Other Study IDs: 0566
Record Dates: First submitted 2016-09-09; First posted 2016-09-26 (Estimated); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Asthma
Keywords: Spirometry; Exhaled Nitric Oxide; Primary Care
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
What are the capacity and training needs in general practice to implement routine spirometry and eNO testing in children aged 5-16 years?

Asthma is the commonest long-term disease of childhood in the United Kingdom (UK). Under-diagnosis and under-treatment of childhood asthma in general practice (GP) have been reported from several European countries including the UK. This can result in poor symptom control and increased risk of asthma related deaths.

It has been suggested that both under- and over- diagnosis of childhood asthma in general practice could be improved by routinely using objective lung function testing for diagnosis and monitoring.

The proposed objective lung function tests (spirometry and exhaled nitric oxide measurements - eNO) are already used routinely in UK hospitals, but are not usually available in general practice where most children are cared for.

Why is it important? - Availability of these tests will help health professionals in general practice to look after children with asthma better, and hopefully improve asthma control.

What will this study achieve? - Though it is believed that providing spirometry and eNO in general practice would be beneficial, there is little data on how this can be achieved. This study will employ both qualitative and quantitative measures in order to evaluate the resources required to implement routine spirometry and eNO testing for children in primary care; and to investigate the impact this would have on diagnosis in children with suspected asthma.

How? - The investigators will work with general practices in and around Leicestershire, UK. Firstly, to identify what the barriers are to implementing these tests, and secondly to train the practices to perform and interpret spirometry and eNO independently in children.

Children with suspected or previously diagnosed asthma will be invited for review and lung function testing. The investigators will record the time it takes to train general practices to perform and interpret spirometry and eNO independently, and the additional clinic capacity required to provide these tests.

ELIGIBILITY:
Inclusion Criteria:

1. On the practice asthma register or
2. Are prescribed regular (on repeat prescription) inhaled corticosteroids including beclometasone, fluticasone and budesonide and also search specifically for 'brands' that are commonly prescribed to include 'clenil', 'seretide', 'symbicort', and 'qvar' or
3. Have been prescribed ≥ 2 Salbutamol MDI's in the last 12 months or
4. Had a documented exacerbation of asthma in the last 12 months
5. Able and willing, in the opinion of the Investigator, to give informed consent

Exclusion Criteria:

1. Children who are unable to perform lung function tests for any reason
2. Children and young people <5 years and >16 years
3. Unable or unwilling, in the opinion of the Investigator, to give informed consent

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients registered to participating general practices in Leicestershire and Northamptonshire
Sampling Method: Non-Probability Sample
Enrollment: 613 (Actual)
Dates: Start 2016-06-01; Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erol Gaillard, PhD MRCPCH, Principal Investigator — National Institute for Health Research, Leicester Respiratory Biomedical Research Unit, University of Leicester
Locations (2):
- United Kingdom (2):
  - Countesthorpe Health Centre, Leicester, Leicestershire
  - Lakeside Surgery, Corby, Northamptonshire

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary care practices based in the the East Midlands, England.
  Recruitment between June 2016 and August 2017
Pre-assignment Details: N/A - single group observational study only
Groups:
- Study Cohort: Participating practices Ten practices participated in this study. They served a population of almost 120,000 people, ranging from ~3500 to 48000 registered patients. Geographically, five of the practices were located in inner-city Leicester, three were in surrounding towns, and two were in village locations.
  Participants Electronic database searches identified 1548 eligible children; 1097 (71%) were on their GPs asthma register, and 451 (29%) were not, but had received asthma medications in the previous 12 months.
  In total 614 children responded to the written invitations and attended clinics held between June 2016 and August 2017; of these, 456 (75%) were on the asthma register. Sixty-three percent of children were recruited in the months of March to August, and the remainder in the months of September to February.
  Written informed consent was obtained from carers of 613 children. One parent refused consent and one parent later withdrew their consent without giving a reason, leaving 612 children in total. The characteristics of recruited children are shown in table 1. Overall, the participation rate was 40% of eligible patients, but ranged from 8% to 59% between practices. The practice recruiting only 8% of eligible children was an outlier, and due in part to recruitment at this practice commencing late into the study and therefore fewer clinics (in relation to the practice size) were set up compared with other practices.
Period: Overall Study
Arm/Group | Study Cohort
Started | 613
Completed | 612
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Written informed consent was obtained from carers of 613 children. One parent refused consent and one parent later withdrew their consent without giving a reason, leaving 612 children in total.
Arm/Group | Study Cohort
Number analyzed (Participants) | 612
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.0 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 280
  Male | 332
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 480
  Ethnicity: Asian | 82
  Ethnicity: Black | 21
  Ethnicity: Mixed | 20
  Ethnicity: Other | 9
Number of children with existing asthma diagnosis [Count of Participants; unit: Participants]
  Asthma Diagnosed Previously (on asthma register) | 456
  Asthma not diagnosed previously (not on asthma register) | 156

OUTCOME MEASURES:

1. Primary Outcome: Time Needed to Perform Paediatric Spirometry and eNO Testing in General Practice
Description: Time (minutes) to perform both spirometry and eNO test in children
Time Frame: 12 months
Population: Spirometry attempted in all 612 children but only successful in 575
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Study Cohort
Number analyzed (Participants) | 575
Minutes
  Time to perform spirometry | 4.3 (1.3)
  Time to perform reversibility test | 3.1 (1.0)
  Time to perform eNO | 2.4 (1.0)

2. Primary Outcome: Number of Children in Whom Usable Spirometry and eNO Data Can be Obtained
Description: Number of children (out of 612) able to perform objective tests
Time Frame: 12 months
Population: Objective tests attempted in all 612 children with consent
Measure: Count of Participants; unit: Participants
Arm/Group | Study Cohort
Number analyzed (Participants) | 612
Participants | 575

3. Secondary Outcome: The Number of Children in Whom a Diagnosis of Asthma Can be Confirmed Using Spirometry and eNO Testing
Description: Number of children in whom an asthma diagnosis could be confirmed on objective testing
Time Frame: 12 months
Population: Spirometry and FeNO data were available from 109 children who had received asthma medications in the previous year
Measure: Count of Participants; unit: Participants
Arm/Group | Study Cohort
Number analyzed (Participants) | 109
Participants | 13

4. Secondary Outcome: Change in Paediatric Asthma Quality of Life Questionnaire Score Measured at Enrolment and 3-6 Months Post-enrollment
Description: Timepoints - Assessed at enrolment and at 3-6 months post enrolment Purpose: The Paediatric Asthma Quality of Life Questionnaire (PAQLQ) was developed to measure the functional problems (physical, emotional and social) that are most troublesome to children with asthma.
  Format: The PAQLQ can be administered by an interviewer or self-administered by the child Content: The PAQLQ contains 23 questions that cover three domains: activity limitation, symptoms, and emotional function Scoring: Children are asked to think about how they have been during the previous week and to respond to each of the 32 questions on a 7-point scale (7 = not bothered at all -
  1 = extremely bothered). The overall PAQLQ score is the mean of all 23 responses and the individual domain scores are the means of the items in those domains. A change in score greater than 0.5 on the 7-point scale can be considered clinically important.
Time Frame: PAQLQ score was assessed at enrolment and then again at 3-6 months post enrolment
Population: Number of children with follow up data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Cohort
Number analyzed (Participants) | 226
units on a scale
  PAQLQ score at baselines | 5.92 (1.06)
  PAQLQ score at follow up | 6.02 (1.04)

5. Secondary Outcome: Change in Child Health Utility 9D Questionnaire Score Measured at Enrolment and at 3-6 Months Post-enrolment
Description: Timepoints - measured at enrolment and at 3-6 months post-enrolment Purpose: The CHU9D is a paediatric generic preference based measure of health related quality of life. It consists of a descriptive system and a set of preference weights, giving utility values for each health state described by the descriptive system, allowing the calculation of quality adjusted life years (QALYs) for use in cost utility analysis.
  Format: Consists of nine dimensions of health-related quality of life, including worry, sadness, pain, tiredness, annoyance, school, sleep, daily routine, and activities. The child completes the questionnaire, or a proxy can complete it for younger children Scoring: Scores can range from -0.1059 (min) to 1 (max); with a score of 1 indicating a "state of perfect health", and a lower score indicating worse health. A minimally important difference (MID) of 0.03 is used to assess the magnitude of mean difference when comparing CHU9D scores.
Time Frame: CHU9D score was assessed at enrolment and then again at 3-6 months post-enrolment.
Population: Number of children with follow up data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Cohort
Number analyzed (Participants) | 226
score on a scale
  CHU9D score at baseline | 0.88 (0.16)
  CHU9D score at follow up | 0.85 (0.18)

6. Other Pre Specified Outcome: The Number of Primary Care Staff Who Found Providing Spirometry and eNO Testing for Children Acceptable After Being Trained
Description: Based on responses to a questionnaire administered at the end of their training using pre-determined responses along a 5-point likert scale.
Time Frame: 12 months
Population: Following training and implementation, 23 (85%) staff members responded to the online feedback questionnaire. Please note: healthcare providers were not considered enrolled within the study but did contribute feedback to this assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Primary Care Healthcare Professionals: Participating practices Ten practices participated in this study. They served a population of almost 120,000 people, ranging from ~3500 to 48000 registered patients. Geographically, five of the practices were located in inner-city Leicester, three were in surrounding towns, and two were in village locations.
  Participants Training was delivered to 27 Practice nurses and health care assistants. No staff had previously had training to perform spirometry or FeNO testing in children.
Arm/Group | Primary Care Healthcare Professionals
Number analyzed (Participants) | 23
Participants | 23

7. Other Pre Specified Outcome: The Number of Participants Who Found Spirometry and eNO Testing Acceptable
Description: Based on responses to a questionnaire administered at the end of their asthma review using pre-determined responses along a 5-point likert scale.
Time Frame: 12 months
Population: Feedback forms were completed by 554 (91%) families
Measure: Count of Participants; unit: Participants
Arm/Group | Study Cohort
Number analyzed (Participants) | 554
Participants | 537

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Study Cohort
All-Cause Mortality (participants affected / at risk) | 0/612
Serious Adverse Events (participants affected / at risk) | 0/612
Other Adverse Events (participants affected / at risk) | 0/612

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-25): https://cdn.clinicaltrials.gov/large-docs/72/NCT02913872/Prot_SAP_000.pdf